CLINICAL TRIAL: NCT06037655
Title: Gemcitabine/Cisplatin Combined With Adebrelimab and Mecapegfilgrastim in Neoadjuvant Treatment of Potentially Resectable Biliary Tract Carcinoma, A Single-arm Study
Brief Title: Chemotherapy Combined With Adebrelimab and Mecapegfilgrastim in Neoadjuvant Treatment of Potentially Resectable BTC
Acronym: Modified
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-BTC-II-002
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Biliary Tract Neoplasms
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): NeoAdjuvant Therapy with Adebrelimab plus Mecapegfilgrastim and Gemcitabine/cisplatin followed by the operation
  Interventions: Drug: Total Neoadjuvant Treatment

INTERVENTIONS:
Drug: Total Neoadjuvant Treatment — Adebrelimab (1200 mg) every three weeks intravenously; Mecapegfilgrastim (6 mg) every three weeks intravenously; Gemcitabine (1000 mg/m2) every three weeks on days 1 and 8 intravenously; Cisplatin (25 mg/m2) every three weeks on days 1 and 8 intravenously

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Gemcitabine/cisplatin combined with Adebrelimab and Mecapegfilgrastim in neoadjuvant treatment of potentially resectable Biliary Tract Neoplasms.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, patients giving written informed consent will undergo a 1-week screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requirements will be receive Gemcitabine/cisplatin combined with Adebrelimab and Mecapegfilgrastim three weeks a cycle, surgery was performed after 4 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age ≥ 18 years，≤ 75 years
* Patients with untreated resectable locally advanced biliary tract cancer (BTC) who are difficult to directly resecte surgically
* Ability to provide written informed consent prior to participation in any study-related procedure
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* At least one, not previously irradiated, measurable lesion according to RECIST (version 1.1).
* Adequate organ function

Exclusion Criteria:

* Diagnosis of mixed ampullary, hepatocellular, and cholangiocarcinoma
* Known history of a serious allergy to any monoclonal antibody
* Any active malignancy prior to the start of treatment
* Active or history of autoimmune disease
* Other acute or chronic conditions, psychiatric disorders, or laboratory abnormalities that may increase the risk of study participation
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-25 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 18 weeks
  ORR is defined as patients achieving clinical complete response (CR) or partial response (PR) according to RECIST v1.1

SECONDARY OUTCOMES:
overall survival (OS) | 2 years
  Overall survival

OTHER OUTCOMES:
Progression free survival (PFS) | 2 years
  PFS is defined as time interval from recruitment to tumor progression or censoring
Pathological Complete Response Rate (pCR) | 18 weeks
  pathological complete response rate
Major Pathological Response Rate (MPR) | 18 weeks
  MPR rate was defined as the percentage of patients who achieved a major pathological response (residual tumor ≤10%)

CONTACTS AND LOCATIONS:
Overall Officials: Xiangcheng Li, Study Chair — The First Affiliated Hospital with Nanjing Medical University; Xiaofeng Chen, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No